CLINICAL TRIAL: NCT03492866
Title: The Efficacy of Topical Gentamycin for the Treatment of Hereditary Hypotrichosis Simplex Caused by Heterozygous Nonsense Mutations in CDSN Encoding Corneodesmosin
Brief Title: Efficacy of Topical Gentamycin for Hereditary Hypotrichosis Simplex Caused by Nonsense Mutations in CDSN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-18-ES-0797-CTIL
Record Dates: First submitted 2018-03-18; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Hereditary Hypotrichosis Simplex
MeSH Terms: conditions — Hypotrichosis simplex | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: Assessing in 8 patients the efficacy of topical gentamycin treatment on 1 side of the scalp by determining the amount of hair loss on the treated versus the untreated side of the scalp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentamicin Sulfate (Active Comparator): All subjects will be treated with topical gentamycin applied twice daily (1 fingertip unit (FTU)) to the right half of the scalp. Total study period: 6 months.
  Interventions: Drug: Gentamicin Sulfate
- No treatment (No Intervention): The medication won't be applied to the left half of the scalp.

INTERVENTIONS:
Drug: Gentamicin Sulfate — Topical treatment of 1 side of the scalp twice daily during 6 months
  Arms: Gentamicin Sulfate

SUMMARY:
The scalp-limited for of hereditary hypotrichosis simplex (HHS; MIM146520) is an autosomal dominant form of non-syndromic alopecia which is caused by heterozygous nonsense mutations in the CDSN gene, encoding corneodesmosin (1). The disease features diffuse gradual scalp hair loss that starts in the middle of the first decade of life and progresses to total alopecia till the third decade of life. Recent studies have shown that aminoglycosides have the potential to induce readthrough of nonsense mutations in human cells.

The aim of this study is to investigate whether topical aminoglycosides (Gentamycin) may be beneficial for the treatment of HHS patients carrying nonsense mutations by inducing readthrough.

The Study goals:

To assess the short and long term efficacy of topical gentamycin for the treatment of hereditary hypotrichosis simplex caused by nonsense heterozygous mutations in CDSN.

The primary end point:

To assess scalp hair growth during study period as compared to baseline. Hair growth will be evaluated during enrollment and every 4 weeks. The secondary end points will be time to regrowth for determining efficacy.

DETAILED DESCRIPTION:
Study design: An open label one arm prospective study designed to evaluate the short and long term efficacy of topical gentamycin for the treatment of 8 patients with hypotrichosis simplex of the scalp.

Patients with hypotrichosis simplex of the scalp carrying a nonsense heterozygous mutation in the CDSN gene, who are eligible to the study based on inclusion/exclusion criteria, will sign the informed consent and will start to apply on the right half of scalp topical Gentamycin twice daily. The medication will not be applied to the left half of the scalp. Other local treatments to the scalp should be avoided during the study period. Daily oral medications are allowed. The patients will undergo general blood examination tests at baseline and every 4 weeks for safety measures. Blood tests include CBC, renal and liver function tests. Gentamycin levels will be assessed every 4 weeks.

Assessments on Visit 1:

Inclusion and exclusion criteria (including verifying normal hearing test at baseline prior to enrollment) Enrollment Baseline lab tests (CBC, renal and liver function tests) Physical exam SALT score Vellus hairs presence Pull test Patients self-assessment scale Photographs

Assessments on Follow up visits (every 4 weeks for a total of 6 months):

Physical exam Local site reactions SALT score Half head assessment Vellus hair presence Pull test Patients self-assessment scale Blood tests (CBC, renal and liver function tests) and gentamycin levels Photographs

Study withdrawal:

Patients with serious side effects of Gentamycin topical treatment such as hearing loss and impaired renal function or other serious side effect that according to the investigator judgment might jeopardize the patient's health. These are unexpected via local application and in the presence of intact skin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypotrichosis simplex of the scalp carrying a nonsense heterozygous mutation in the CDSN gene
2. Patients 18 years of age or older
3. Patient with normal hearing assessment within 30 days prior to treatment with the investigational drug
4. Patients with normal liver and renal function

Exclusion Criteria:

1. Patients with Hypotrichosis simplex of the scalp with no identified mutation in CDSN
2. Patients under 18 years of age
3. Patients with known hearing loss and renal and liver insufficiency
4. Patients with impaired skin barrier over the scalp such as bruise, ulcer, erosion etc.
5. Pregnancy and breastfeeding

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Hair density over the scalp | During 6 months of treatment
  The Severity of Alopecia Tool (SALT) Score will be the measure of hair density as following: Percentage of terminal hair loss is determined at the top of the scalp (A), the back of the scalp (B), left side of the scalp (C) and right side of the scalp (D). The sum of A+B+C+D = SALT score.

SECONDARY OUTCOMES:
The presence of vellus hairs | During 6 months of treatment
  The appearance of vellus hair on the treated half scalp versus the untreated half scalp is a qualitative measure for Gentamycin efficacy
Activity of hair loss | During 6 months of treatment
  The hair pull test will indicate if active hair loss is present or not, in the treated half of the scalp versus the untreated half of the scalp as a measure for Gentamycin efficacy
Photographic documentation | During 6 months of treatment
  Pictures of the scalp will be taken to illustrate Gentamycin effect
Side effects | During 6 months of treatment
  Patients will be asked if they experienced side effects of topical Gentamycin treatment: local site reactions such as erythema, , irritation, dryness

CONTACTS AND LOCATIONS:
Overall Officials: Liat Samuelov, Study Director — Deprt. of Dermatology, Tel Aviv Sourasky MC